CLINICAL TRIAL: NCT01885468
Title: X-Ray Verified Accuracy of the Aesculap - Miethke proGAV Adjustable Shunt Pressure Setting Verification Instrument
Brief Title: X-Ray Verified Accuracy of the proGAV Verification Instrument
Acronym: X-AMIN
Status: Completed | Type: Observational
Sponsor: Aesculap, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: AAG-G-H-1106
Record Dates: First submitted 2013-06-21; First posted 2013-06-25 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2017-01

CONDITIONS: Hydrocephalus Shunt (proGAV) Requiring Adjustment
Keywords: Hydrocephalus shunt; proGAV

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is to verify the use of a hand held tool to verify the new setting of a hydrocephalus shunt (proGAV). This tool would be used in place of an Xray of the patient's head, which is how settings are verified currently.

ELIGIBILITY:
Inclusion Criteria:

* Implanted with proGAV Requiring adjustment Implant must be palpable under the skin

Exclusion Criteria:

* Unwilling to consent Implanted within 7 days of inclusion visit

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hydrocephalus patients implanted with proGAV shunt requiring adjustment
Sampling Method: Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2013-05; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Level of agreement between the proGAV® verification instrument measurement and X-ray control measurements. | 1day

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Valley Children's Hospital, Madeira, California
  - Geisinger Medical Center, Danville, Pennsylvania